CLINICAL TRIAL: NCT02215109
Title: Change of Retinal Vessel Diameter in Branch Retinal Vein Occlusion After Intravitreal Bevacizumab Injection
Brief Title: Retinal Vessel Diameter in Branch Retinal Vein Occlusion
Status: Completed | Type: Observational
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Dong Ho Park, Clinical professor, Kyungpook National University Hospital
Other Study IDs: KNUHOPH2014-01
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Branch Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- BRVO, Retinal vessel diameter: The retinal vessel diameter was measured Branch Retinal Vein Occlusion patients after intravitreal bevacizumab injection.

SUMMARY:
The authors investigated the consecutive change of retinal vessel's diameter in affected eye and fellow eye of Branch Retinal Vein Occlusion.

DETAILED DESCRIPTION:
Twenty five consecutive patients who had undergone intravitreal bevacizumab injection for Branch Retinal Vein Occlusion with macular edema were included in this study. All subjects were enrolled between April, 2012 and April, 2013 in the Department of Ophthalmology, Kyungpook National University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Best-corrected visual acuity less than 20/40
* Central subfield macular thickness (CSMT) 300 μm or greater on spectral-domain optical coherence tomography

Exclusion Criteria:

* Patients with recurrent BRVO
* History of previous treatments for BRVO including vitreoretinal surgery, intravitreal injection, subtenon injection or laser photocoagulation
* Patients with diabetes or dyslipidemia
* IOP ≥ 22mmHg, treatment for glaucoma, a family history of glaucoma, or optic neuropathy
* High myopia (<-6 Diopters), high hyperopia (>6 Diopters) or a history of refractive surgeries
* Co-existing retinal disease other than BRVO
* Corneal diseases include ulcer, keratoconus and a history of corneal laceration
* Cataract and other media opacities resulting in visual impairment or poor fundus images

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 25 patients will be included. All subjects with branch retinal vein occlusion scheduled for intravitreal bevacizumab injection.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-04; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Unoccluded retinal vessel diameter of Branch Retinal Vein Occlusion | 0, 1, 3, and 6 months
  To evaluate the change of unoccluded retinal vessel diameter in affected eye of Branch Retinal Vein Occlusion and unaffected fellow eye.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ho Park, M.D., Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Dong Ho Park, Daegu, Kyungsangpookdo, South Korea

IPD SHARING:
Plan to Share IPD: No